CLINICAL TRIAL: NCT06857604
Title: The Interplay Between Inborn Error of Immunity and Blood Disorders: Unravelling Immune Defects Behind Common Haematological Diseases
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meyer Children's Hospital IRCCS (Other)
Responsible Party: Principal Investigator, Eleonora Gambineri, Medical Doctor, Meyer Children's Hospital IRCCS
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IEI-Haem
Record Dates: First submitted 2025-02-24; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Hematologic Diseases
MeSH Terms: conditions — Hematologic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients with Haematological Disorders (Other): Patients with diagnosed autoimmune cytopenias (AIC), polyclonal lymphoproliferation (PL), lymphoma (ML), bone marrow failure, and myelodysplastic syndrome (BMF/MDS)
  Interventions: Other: Biological samples

INTERVENTIONS:
Other: Biological samples — Immunological Screening and Genetic analysis

SUMMARY:
The universe of Inborn errors of Immunity (IEI) is rapidly expanding: their clinical spectrum is not only characterised by infections but often includes haematological complications. Moreover, an increasing number of "IEI phenocopies" due to somatic mutations in specific cell types are progressively being unveiled and complicate the genetic plot of IEI, which are therefore not only caused by germline mutations. However, these aspects have never been studied by large prospective studies.

This study aims to fill this gap by prospectively recruiting patients <25 y/o with haematologic disorders that fall into one of the following 4 subgroups: autoimmune cytopenia (AICs), polyclonal lymphoproliferation (PL), monoclonal (malignant) lymphoproliferation (ML), bone marrow failure/myelodysplasia (BMF/MDS). Recruited subjects will undergo an extensive immunologic workup (extended immunophenotyping, cytokine and autoantibody dosage) together with genetic testing (NGS) to detect both germline and somatic variants. Bulk RNA sequencing will be performed either as functional validation of variants or to identify altered pathways in selected cases with inconclusive genetics. Patient advocacy organisations (PAOs) will be pivotal to assist patients' needs throughout the project and to raise awareness of predictive and yet unknown signs of IEI.

The study involves recruitment a total of almost 700 children over a 3-year period. Considering recent studies on AICs and BMF/MDS, a global detection rate of 30% "hidden" IEI is expected, with higher rates in the AIC subgroup and lower ones for ML, given the complexity of lymphoma pathogenesis. New IEI candidate genes or new examples of IEI phenocopies are expected to be identified.

The immunological workup should detect early disease biomarkers or currently unknown molecular signatures of specific disorders. These may increase the chance of identifying an IEI in a specific subgroup and promptly address the patient to a targeted treatment or to hematopoietic stem cell transplantation, avoiding late complications, increasing patients' survival, and abating the economic burden of the disease on healthcare services. Finally, involvement of PAOs may foster patients' knowledge about their condition, increasing their compliance to disease follow-up and treatment and ameliorating their quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age < 25 years
2. Patients with diagnosed autoimmune cytopenias (AIC), polyclonal lymphoproliferation (PL), lymphoma (ML), bone marrow failure, and myelodysplastic syndrome (BMF/MDS) (see details below)
3. Signed Informed Consent

Exclusion Criteria:

1. Patients with Lymphoma secondary to HIV or transplant
2. Patient with self-resolving or post-infective AICs

Max Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 700 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Number of children and young adults with blood disorders with new or known germline and somatic mutations that cause or modify disease, either in the lymphoid or myeloid compartments. | From enrollment to the end of analysis (36 months)

SECONDARY OUTCOMES:
Percentage of pediatric and adolescent-young adult patients with hematologic disorders with altered immunological profiles | From enrollment to the end of analysis (36 months)

CONTACTS AND LOCATIONS:
Locations (6):
- CHU Sainte-Justine, Montreal, Canada, Canada
- Institut Imagine, Paris, France, France
- Italy (2):
  - Meyer Children's Hospital IRCCS, Firenze, Florence, Fi
  - University of Rome Tor Vergata, Rome, Italy
- Vall d'Hebron Institut de Recerca, Barcelona, Spain
- Karolinska Institutet, Stockholm, Sweden, Sweden

IPD SHARING:
Plan to Share IPD: No